CLINICAL TRIAL: NCT07033546
Title: The Effect of Using Toy Bracelets During Physical Restraint in a Pediatric Intensive Care Unit on Children's Physiological Parameters, Fear, and Anxiety Levels: A Randomized Controlled Trial
Brief Title: The Effect of Using Toy Bracelets During Physical Restraint in a Pediatric Intensive Care Unit on Children's Physiological Parameters, Fear, and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OKAN_UNV
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Intensive Care Unit; Physical Restraint; Anxiety; Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental)
  Interventions: Behavioral: Toy bracelets

INTERVENTIONS:
Behavioral: Toy bracelets — The intervention involves the use of colorful, child-friendly toy bracelets worn by children during procedures requiring physical restraint in the pediatric intensive care unit. These bracelets are designed to offer a sense of familiarity, distraction, and emotional comfort during potentially distressing experiences. Unlike standard care, which involves restraint without any therapeutic distraction tools, the toy bracelets serve as a non-pharmacological, low-cost, and easily applicable intervention aimed at reducing emotional distress. The intervention is distinguished by its simplicity, immediate usability, and focus on integrating play-based elements into clinical care to address the psychological needs of hospitalized children.
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aimed to evaluate the effects of using toy bracelets during physical restraint on physiological parameters, fear, and anxiety levels in children aged 4 to 12 years in a pediatric intensive care unit. Conducted between December 2023 and December 2024 at Istanbul Şehit Prof. Dr. İlhan Varank Training and Research Hospital, the study included 65 children, with 32 in the intervention group and 33 in the control group. Data collection tools included the Child Information Form, Child Fear Scale, and State-Trait Anxiety Inventory for Children (STAI-C), along with calibrated devices for physiological monitoring. Assessments were carried out at baseline and during the first, second, and third hours of observation to evaluate the intervention's impact over time.

ELIGIBILITY:
Inclusion Criteria

* Children aged between 4 and 12 years
* Child is conscious
* First admission to the intensive care unit
* First-time experience of physical restraint
* Parental consent for the child's participation in the study

Exclusion Criteria

* Intubated patients
* Presence of burns, wounds, or similar conditions on the limb to be restrained
* Hearing impairment
* Known mental illness
* Deep sedation administered (exceeding ketamine 1 mg/kg or midazolam 0.5 mg/kg)
* Presence or suspicion of cranial or any other type of bleeding
* Neurological disorder
* Terminal stage of illness

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Children Fear Scale | Fear was assessed at baseline and at the first, second, and third hours after admission of the children.
  The Child Fear Scale consists of six facial expressions scored from 0 (no fear) to 10 (highest fear) in increments of two. Fear increases progressively across the faces. Its validity and reliability were confirmed by Avşan et al. (2024), and it aligns with pain scales in format and scoring.
Child Anxiety State Scale | Anxiety was assessed at baseline and at the first, second, and third hours after admission of the children.
  The Child Anxiety State Scale (CAS-S), developed by Ersig et al. (2013), was validated in Turkish by Özalp Gerçeker et al. (2019). Designed for children aged 4-10, it resembles a thermometer and measures current anxiety ("right now"). The scale has strong psychometric properties and is suitable for clinical use.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No